CLINICAL TRIAL: NCT04680845
Title: INSPIRES Hearing Health Trial - INnovative Psychological Intervention to REduce Stigma in Hearing Health Trial
Acronym: INSPIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Christopher Armitage, Professor of Health Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-10597-17109
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-affirmation (Experimental): Participants will be asked to complete a standard questionnaire including:
  The beginning to a sentence appears below. Below it are 4 different ways of completing the sentence. On the lines below, please write out the beginning of the sentence and then complete it with 1 of the 4 options we have given you.
  If I feel threatened or anxious, then I will… …think about the things I value about myself
  * remember things that I have succeeded in
  * think about what I stand for
  * think about things that are important to me
  If…______________________________________________________________________
  Interventions: Behavioral: Self-affirmation
- Control (No Intervention): Participants will be asked to complete a standard questionnaire.

INTERVENTIONS:
Behavioral: Self-affirmation — According to self-affirmation theory (Steele, 1988), defensiveness arises because people are motivated to defend their global sense of self-worth, which in the present case is threatened by perceptions of hearing aids/loss. However, if a person's self-image can be bolstered (affirmed) in a domain that is important to them, thereby preserving self-integrity, the individual should be less likely to process the threatening (i.e., stigmatizing in the present context) information defensively (Steele, 1988).
  Arms: Self-affirmation

SUMMARY:
Background: Reminding people they are moral adaptable human beings ("self-affirming") reduces the perceived stigma associated with wearing hearing aids and increases actual hearing aid use. The proposed study aims to reduce stigma in a representative sample of people aged over 60 from the general population who may or may not already be wearing hearing aids and improve multiple hearing health outcomes (e.g., attending screening, device use).

Methods/Design: Double-blinded randomized controlled trial in which a representative sample of people aged over 60 from the general population will be asked to complete surveys about hearing stigma, hearing loss and multiple hearing health outcomes. Participants randomized to the control group will only complete the survey; participants in the intervention group will be asked to affirm their values. Six months later, all participants will complete the same survey to assess outcomes.

Discussion: The proposed research will lead to a brief psychological intervention to reduce stigma in relation to hearing loss/aids.

DETAILED DESCRIPTION:
According to self-affirmation theory, defensiveness arises because people are motivated to defend their global sense of self-worth, which in the present case is threatened by perceptions of hearing aids/loss. However, if a person's self-image can be bolstered (affirmed) in a domain that is important to them, thereby preserving self-integrity, the individual should be less likely to process the threatening (i.e., stigmatizing in the present context) information defensively. Accumulated empirical evidence demonstrates that affirming the self: (a) reduces public stigma, (b) reduces self-stigma, and (c) causes meaningful changes in behaviour. Following a pilot-feasibility trial showing that self-affirming caused significant reductions in first-time hearing aid users' anxieties about ageing and increased their hearing aid use by almost 2 hours/day.

ELIGIBILITY:
Inclusion Criteria:

* UK-based adults
* Aged 60+

Exclusion Criteria:

* Adults younger than 60 years
* Not UK-based

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3012 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Hearing loss public stigma | 6 months
  Self-report questionnaire comprising seven items on 7-point Likert-type scales where 1 = low stigma and 7 = high stigma
Hearing aid public stigma | 6 months
  Self-report questionnaire comprising seven items on 7-point Likert-type scales where 1 = low stigma and 7 = high stigma
Hearing loss self-stigma | 6 months
  Self-report questionnaire comprising five items on 7-point Likert-type scales where 1 = low stigma and 7 = high stigma
Hearing aid self-stigma | 6 months
  Self-report questionnaire comprising nine items on 7-point Likert-type scales where 1 = low stigma and 7 = high stigma

SECONDARY OUTCOMES:
Hearing health seeking behaviours | 6 months
  Self-report questionnaire comprising eighteen items on no-yes scales where 0 = "no" and 1 = "yes"
Spontaneous self-affirmation | 6 months
  Self-report questionnaire comprising two items on 4-point Likert-type scales where 1 = low spontaneous self-affirmation and 4 = high spontaneous self-affirmation
Subjective well-being | 6 months
  Self-report questionnaire comprising four items on 11-point Likert-type scales where 0 = low subjective well-being and 10 = high subjective well-being
Anxiety about ageing | 6 months
  Self-report questionnaire comprising three items on 7-point Likert-type scales where 1 = low anxiety and 7 = high anxiety

OTHER OUTCOMES:
Impact of Covid-19 | 6 months
  Self-report questionnaire comprising fifteen items on 4-point Likert-type scales where 1 = low impact and 4 = high impact

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Munro, PhD, Study Chair — University of Manchester
Locations (1):
- YouGov, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The dataset used during the current study are available from the research team on reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Following publication of the main paper for 5 years.
Access Criteria: On reasonable request.